CLINICAL TRIAL: NCT04436055
Title: Intergenerational Effects of Paternal Periconceptional Cannabis and Other Drug Use (EPIC)
Acronym: EPIC
Status: Terminated | Type: Observational
Why Stopped: Sponsor did not renew funding.
Sponsor: Duke University (Other)
Collaborators: John Templeton Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00105659
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2022-04

CONDITIONS: Cannabis Use; Drug Use; Development, Infant

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants: All participants including cannabis users, other drug users, and non-drug users.
  Interventions: Other: No Intervention will be used

INTERVENTIONS:
Other: No Intervention will be used — Since this is an observational study, there are no interventions.

SUMMARY:
The overall objective of this proposed project is to prospectively evaluate the epigenetic and developmental effects of paternal cannabis and other drug use in offspring.

DETAILED DESCRIPTION:
This project involves enrollment of 40 healthy mother-father dyads that are between the ages of 18 and 40 years. Urine samples for qualitative drug and cotinine testing will be collected from mother-father dyads, as well as quantitative THC (tetrahydrocannabinol) and THCCOOH (11-nor-9-carboxy-THC) assay. A semen sample will be collected from biological fathers. Relevant birth outcome data including both infant and maternal measures will be extracted from the electronic health record (EHR). Infant developmental assessments will be completed at approximately 6 months of age.

ELIGIBILITY:
Inclusion Criteria:

1. Both mother and father are between 18 and 40 years of age
2. Free from significant medical conditions, as determined by medical history and examination from attending Obstetrician or health care provider.
3. Father is able to be contacted and consents to provide urine and sperm samples
4. Both mother and father consent to participation and for the prospective enrollment of their child after birth
5. Plan on delivering their baby at one of the two main Duke-affiliated hospitals (Duke University Medical Center and Duke Regional Hospital)

Exclusion Criteria:

1. Mother or Father currently prescribed any psychoactive medication;
2. Mother or Father unable to comply with study requirements or otherwise unsuitable for participation in the opinion of the PI.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 40 mother-father dyads.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Methylation profiles for fathers and offspring | Intake visit for fathers; 6 months after birth for offspring
  Examine methylation profiles from fathers with varying patterns of drug use as well as from fathers with no drug use; and determine whether methylation profiles are transmitted to offspring.
Extent to which cannabis and other drug related epigenetic effects in fathers are associated with birth outcomes in offspring | Intake visit for fathers; 0-6 months for offspring
  Electronic health record data will be used to assess a range of perinatal outcomes in babies and evaluate their association with paternal drug use status and accompanying methylation profiles in fathers and offspring.
Differences in developmental functioning in babies born to fathers using cannabis and other drugs; and to explore whether any observed differences are mediated by differences in methylation profiles of offspring saliva cells. | Intake visit for fathers; 6 months for offspring
  Developmental functioning in babies will be assessed at approximately 6 months of age and their association with paternal drug use status and accompanying methylation profiles in fathers and offspring will be evaluated. .

CONTACTS AND LOCATIONS:
Overall Officials: John Mitchell, PhD, Principal Investigator — Duke University; Tiffany Covas, MD, Principal Investigator — Duke University
Locations (1):
- Duke Child and Family Study Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No